CLINICAL TRIAL: NCT00445523
Title: A Phase II Trial to Assess the Activity of TroVax® Alone vs. TroVax® Plus Interferon Alfa (IFN-α) on Patients With Advanced or Metastatic Renal Cell Cancer
Brief Title: Safety Study of TroVax Alone vs. TroVax Plus Interferon Alpha in Patients With Renal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0206-0028; TV2/002/06
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Advanced renal cancer; metastatic renal cancer; RCC; kidney cancer; M3thodist
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — TroVax; Interferon-alpha; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): TroVax® alone
  Interventions: Biological: TroVax® (Immunological Vaccine Therapy)
- 2 (Experimental): TroVax® plus IFN-α
  Interventions: Biological: TroVax® (Immunological Vaccine Therapy); Drug: Interferon-alpha

INTERVENTIONS:
Biological: TroVax® (Immunological Vaccine Therapy) — 16 Intramuscular injections of TroVax® over 47 weeks
Drug: Interferon-alpha — 36 subcutaneous IFN-α injections for 12 weeks. sc injection three times per week (5MU each)
  Other Names: Intron
  Arms: 2

SUMMARY:
Patients with metastatic renal cell cancer will be enrolled to receive either Trovax® alone or Trovax® plus Interferon Alfa. The study will try to determine whether the use of Trovax® will delay tumor progression.

DETAILED DESCRIPTION:
Patients with metastatic renal cell cancer will be enrolled in the study if all inclusion/exclusion criteria are met. Once the patient is enrolled, and baseline tests have been completed, the patient will start treatment.

Trovax® alone arm:

Trovax will be given as an intramuscular injection every two weeks for the first two months, then once a month for the next 2 months, and then once every 2 months for up to a year.

Trovax® plus IFN-α:

Trovax® schedule will be the same as the Trovax® alone arm. IFN will be given on the first, third and fifth day of the week for a total of twelve weeks.

At every office visit vital signs will be taken. Every eight weeks a medical history, physical exam, performance status evaluation, chest x-ray or CT scan, abdomen/pelvis CT scan or MRI will be done. A blood sample (about 8-10 tablespoons) will be taken to test the immunological response to TroVax® on the same days that the patient receives TroVax® injections.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic histologically confirmed clear cell or papillary cell renal carcinoma.
* Primary tumor surgically removed.
* Stable or progressive disease as defined by RECIST criteria.
* Age ≥ 18 years.
* At least one prior standard of care therapy (IL-2, IFN-α, or approved kinase inhibitor)
* At least four weeks from prior use of standard of care therapy.
* Karnofsky performance status ≥ 80%.
* Corrected Serum Calcium ≥ 10 g/dL.
* Patients on stable doses of bisphosphonates (Fosamax, Actonel, Didrocal) that show subsequent tumor progression may continue on this medication; however patients are not allowed to start bisphosphonates within one month prior to starting trial, or throughout the duration of the trial.
* Major surgery or radiation therapy completed ≥ 4 weeks prior to treatment.
* Clinically immunocompetent.
* Free of clinically apparent autoimmune disease.
* Absolute lymphocyte count ≥ 500/μL, Absolute neutrophil count ≥ 1200/μL, Platelet count ≥ 100,000/μl, Hemoglobin ≥ 9mg/dL.
* No evidence of active ischemia on Electrocardiogram (ECG)
* Women must be either post-menopausal, rendered surgically sterile, or using reliable form of contraceptive.
* Able to give informed consent and comply with the protocol.

Exclusion Criteria:

* Prior treatment with TroVax®
* No supplements of complementary medicines/botanicals are permitted during study, except for any combination of the following: multivitamins, selenium, lycopene, soy supplements, Vitamin E.
* Prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
* Participation in any other clinical trial within 30 days.
* Cerebral metastasis on MRI Scan.
* Currently active second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse.
* Serious intercurrent infections or nonmalignant medical illnesses which are uncontrolled.
* Psychiatric illnesses that would limit compliance with protocol.
* A history of psychosis or clinical depression.
* Liver function tests (ALT, AST) more than 1.5 X upper limit of normal (ULN). Bilirubin must be within normal limits.
* Creatinine ≥ 1.5 X ULN.
* Known allergy to egg proteins.
* Known allergy to neomycin.
* History of allergic response to previous vaccinia vaccinations.
* Chronic oral corticosteroid use unless prescribed as replacement therapy in the case of adrenal insufficiency.
* Positive for HIV or Hepatitis B or C.
* Clinical indication of reduced cardiac function or an ejection fraction of ≤ 40%.
* Pregnancy or lactation
* Current chemotherapy, immunotherapy, radiation therapy, or the requirement for radiotherapy.
* No investigational or commercial agents or therapies other that those included in the protocol treatment may be administered with the intent to treat malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-05; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Tumor objective response rate by RECIST criteria to TroVax® and TroVax® in combination with IFN-α. | restaging every 9 weeks

SECONDARY OUTCOMES:
Overall survival | restaging every 9 weeks
Progression-free survival | restaging every 9 weeks
Time to Progression | restaging every 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No